CLINICAL TRIAL: NCT01595334
Title: Is it Possible to Obtain Higher Yield of Mature M2 Oocytes by Establishing Appropriate Levels of LH During Controlled Ovarian Hyperstimulation (COH) in Antagonist Cycles for In-vitro Fertilization-embryo Transfer (IVF-ET)/ Intracytoplasmic Sperm Injection (ICSI)?
Brief Title: Study on Influence of Leutinizing Hormone (LH) on Oocyte Maturity
Acronym: LH/M2-Oocyte
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Cross Fertility Centre (Other)
Collaborators: Disha Fertility and Surgical Centre,Indore,India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB/LH-M2/OM/2011
Record Dates: First submitted 2012-04-27; First posted 2012-05-10 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Infertility
Keywords: IVF-ET; ICSI; Gonadotrophins; rFSH; rLH; Cetrorelix; Leuprolide acetate
MeSH Terms: conditions — Infertility | interventions — cetrorelix; luprolide acetate gel depot; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study subjects desiring pregnancy (Active Comparator): Study subjects to be treated with rFSH, rLH throughout controlled ovarian hyperstimulation (COH) in appropriate dosages,considering age, body mass index (BMI), ovarian reserve, etc. and GnRH antagonist, cetrorelix in 0.25 mg/d when needed till the desired follicular maturity and the minimum required number of follicles are achieved.
  INTRVENTIONS - Monitoring at regular intervals by transvaginal ultrasound and hormonal studies.Once pregnancy established by beta-human chorionic gonadotropin (hCG) and ultrasound will be supported by intervention of adequate luteal support by estrogen (E) + progesterone (P) for 12 weeks of gestation.
  Interventions: Drug: Cetrorelix
- Control subjects desiring pregnancy (Other): Control subjects selected in randomized way,desiring pregnancy will be treated with gonadotrophins, rFSH and rLH in appropriate dosages considering age, BMI, ovarian reserve, etc. after standard downregulation with GnRH agonist, Leuprolide acetate, 1 mg/d under established 'Long Luteal Suppression Protocol' from the previous cycle.
  INTERVENTIONS - Monitoring of response to treatment by hormonal study and sonography evaluation at regular intervals during COH till adequate number of mature follicles of minimum 18 mm mean diameter is achieved, to be followed by hCG trigger and ovum pick-up (OPU) and embryo transfer (ET). Chemical pregnancy by beta-hCG would be confirmed 14 days post-ET. Clinical pregnancy would be confirmed by sonography 6 weeks after ET (visibility of yolk sac and fetal heart-beat). Pregnancy support by E+P for 12 weeks would be provided.
  Interventions: Drug: Luprolide Acetate

INTERVENTIONS:
Drug: Cetrorelix — Cetrorelix 0.25 mg/d would be administered by subcutaneous injection to women when the plasma LH is higher (>4.5 mIU/ml) in the study arm
  Other Names: Cetrotide
  Arms: Study subjects desiring pregnancy
Drug: Luprolide Acetate — Women in the control arm would receive Luprolide acetate 1 mg/day by subcutaneous injection
  Other Names: Lupron
  Arms: Control subjects desiring pregnancy

SUMMARY:
1. Leutinizing hormone (LH) has been demonstrated to exert variable physiological actions during menstrual cycle at appropriate plasma levels'
2. In early follicular phase,in the requisite range,LH is known to contribute to maturation of oocyte during transition phase from metaphase-1(M1) to metaphase-2 (M2).
3. If during this transition, appropriate level of LH can be maintained either through the use of gonadotropin releasing hormone (GnRH) antagonist if found excessive or supplementation with exogenous LH, if found deficient, maturation process can be enhanced.
4. Further maintenance of suitable combination of recombinant follicle stimulating hormone (rFSH) + rLH can help in realizing higher yield of mature M2 oocytes,with higher probability of establishing clinical pregnancy.

DETAILED DESCRIPTION:
The study is planned to assess whether maintenance of levels of LH through the use of GnRH antagonist would contribute to obtaining mature M2 oocytes so that maximum number of good quality embryo's with potential to implant is obtained.

The mature oocytes would be subjected to either standard in-vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) depending on the status of the male factor.

The objective would be to obtain good quality embryo's with implantation potential for fresh embryo transfer and/or subsequent frozen thaw embryo transfer.

In both these events, the secondary outcome measures would be establishment of clinical pregnancy by transvaginal ultrasound performed 6 weeks after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years
* Primary or secondary infertility
* Desire to achieve pregnancy
* Basal FSH <12 mIU/ML
* Moderate to good ovarian reserve (antimullerian hormone (AMH) >1ng/ml, and/ or antral follicle count (AFC)>8 between both ovaries)
* Informed written consent from both partners
* BMI <35 kg/mtr.sq.
* No genetic abnormality

Exclusion Criteria:

* Hormonal preparation taken within 3 month prior to recruitment
* Women with previous poor response to gonadotrophins
* History of previous 3 or more miscarriages
* Women with uncorrected tubal/uterine pathology
* Women opting for assisted procedures like embryo hatching etc.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-09 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Number of mature oocytes immediately after oocyte recovery | Women would be followed every 2 weeks upto 6 weeks after embryo transfer
  Number of mature oocytes would be measured immediately after the oocyte recovery

SECONDARY OUTCOMES:
Clinical pregnancy | Women would be followed every 2 weeks upto 6 weeks after embryo transfer
  Diagnosed by transvaginal ultrasound.Appearance of yolk sac with fetal heart beat at 6 weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: M R Bharucha, PhD, Study Director — Sat Kaival Pvt. Ltd, Anand, Gujarat; Nayana Patel, MD, Principal Investigator — Sat Kaival Hospital Pvt. Ltd, Anand, Guajarat; Faram Irani, MD, Principal Investigator — Southern Cross Fertility Center, Mumbai, India; Asha Baxi, MD, FRCOG, Principal Investigator — Disha Fertility & Surgical Hospital, Indore, India
Locations (3):
- India (3):
  - Sat Kaival Hospital Pvt. Ltd., Anand, Gujarat
  - Disha Fertility & Surgical Hospital, Indore, Madhya Pradesh
  - Southern Cross Fertility Center, Mumbai, Maharashtra